CLINICAL TRIAL: NCT02804789
Title: European Prevention of Alzheimer's Dementia (EPAD) Longitudinal Cohort Study (LCS)
Acronym: EPAD-LCS
Status: Terminated | Type: Observational
Why Stopped: No further funding available, remaining visits halted due to threat of Covid 19
Sponsor: University of Edinburgh (Other)
Collaborators: Innovative Medicines Initiative (Other)
Responsible Party: Sponsor
Other Study IDs: EPAD-UoE-001
Record Dates: First submitted 2016-05-09; First posted 2016-06-17 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Alzheimer's Dementia
Keywords: Prevention
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 44 Months
Biospecimen Retention: Samples With DNA — * Urine
  * Saliva
  * CSF
  * Blood (Serum, Plasma, Whole Blood, RNA, DNA)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Brain changes associated with Alzheimer's disease may precede symptoms of Alzheimer's Dementia by over 20 years. The Investigators hope to be able to identify Alzheimer's disease at its very earliest stages when in theory treatments are most likely to be successful in preventing further spread of the disease in the brain and causing dementia. The aim of EPAD programme is to develop new treatments more quickly to prevent Alzheimer's dementia. A major component of the EPAD programme is the EPAD Longitudinal Cohort Study which can provide subjects for the EPAD trial as well as data to improve understanding of disease before dementia develops.

The Investigators will approach a broad range of people over the age of 50 who have previously taken part in various research studies and consented to being recontacted for further research. Participants will be asked questions to assess their memory and other cognitive function. The participants will also undertake a brain scan, provide a sample of spinal fluid, blood, urine and saliva to look at markers in these bodily fluids that may change in Alzheimer's disease. The Investigators will then follow these participants until December 2019 repeating these tests annually. This will be called the EPAD Longitudinal Cohort Study (EPAD LCS). The main reasons for EPAD developing a cohort are to help the Investigators understand more about what happens to people before dementia develops, and to help recruit people more quickly into the EPAD trials of new medications or other interventions expected to prevent dementia.

People in the EPAD LCS may be invited to take part in the EPAD Proof of Concept prevention studies to see if interventions can modify the probability of developing dementia or cognitive problems (this will be subject to separate ethics approval and consent). Together EPAD LCS and EPAD PoC make up the full EPAD Programme.

DETAILED DESCRIPTION:
The EPAD project has been established to overcome the major hurdles hampering drug development for secondary prevention of AD dementia, by conducting the EPAD LCS (fed mainly from existing Parent Cohorts (PC) across Europe) in alignment with the adaptive design EPAD PoC trial. Both EPAD LCS and EPAD PoC trial will be run in an exclusive network of highly selected, expert Trial Delivery Centres (TDC) that will be selected on the basis of strictly applied criteria to ensure the highest possible data quality, successful recruitment and adherence to the EPAD principles.

While interventions must start early in the course of AD, accurate disease models covering the entire course of AD before dementia onset are lacking. Estimating with reasonable confidence an individual's overall probability of developing AD dementia over a defined time period must take into account multiple dimensions simultaneously (e.g. cognition, biomarkers, traditional risk factors - genetic and environmental). This will allow any given individual to be placed somewhere on a probability spectrum from negligible probability to high probability. Because individuals with similar overall probability may have very different contributions from various components in each dimension, flexible algorithms are needed instead of simple cut-offs to identify a probability-spectrum population adequate for both disease modelling and for providing a sufficient number of potential trial participants (especially in adaptive trials with multiple arms testing drugs with different mechanisms of action).

EPAD LCS is designed to address the dual need for development of accurate longitudinal models for AD covering the entire disease course, and development of adequate infrastructure for facilitating identification of research participants and clinical trial recruitment. EPAD LCS will have a probability-spectrum population selected mostly from already existing PCs across Europe to facilitate fast recruitment. Different types of PCs will be considered (e.g. memory clinic-based, population-based). Due to the variety of PCs, some EPAD LCS research participants will be e.g. memory clinic patients without dementia, while others will be e.g. participants without dementia from the general population. The variety of PC settings will ensure that the EPAD LCS probability-spectrum population can cover the entire continuum of probability for AD dementia development. Regular EPAD LCS follow-up with clinical, cognitive and biomarker assessments will provide a well-phenotyped probability-spectrum population, generating high-quality data for updating disease models, for easier identification of individuals suitable for trial inclusion, and for use as trial run-in data and reference for evaluating intervention efficacy.

The flow of research participants from the population at large to the trial is divided into the following stages: firstly, EPAD will engage existing PCs from across Europe who may have eligible research participants for the EPAD LCS. The next step is drawing research participants from the PCs into the EPAD LCS to maintain a suitable population of approximately 6,000 research participants. Recruitment will be complemented with research participants who are recruited from a clinical setting by their referring clinician. To enable access to the EPAD LCS for these potential participants, the referring clinician will check if they match the flexible algorithm. Finally, research participants in the EPAD LCS who fulfil trial inclusion criteria (approximately 1,500 research participants), will be invited to enter the EPAD PoC (PoC) trial for evaluation of treatment for secondary prevention of AD dementia. This trial is a standing, adaptive, PoC trial that could involve multiple arms running concurrently. Successful graduation through PoC into phase 3 confirmatory trials of single or combinatorial interventions will be based on success against an intermediary, target specific biomarker and then success against a cognitive measure.

Once recruitment is completed, at any given time there should be approx. 6,000 research participants in the EPAD LCS and approx. 1,500 in the EPAD PoC, hence the need to replenish each from PCs as participants are lost through attrition. EPAD LCS will initially run until the end of December 2019, and extension of consent will be sought after 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. At least 50 Years of Age
2. Characterisation of cognitive, biomarker and risk factors (genetic, environmental) status of research participants based on data collected at the EPAD screening/baseline visit, so that decisions on selection/deselection can be made with reference to the dual needs of having sufficient heterogeneity across the entire probability-spectrum population for disease-modelling work, and suitable research participants for the EPAD PoC trial (Balancing Committee decision)
3. Able to read and write with a minimum of 7 years of formal education.
4. Willing in principle to participate in the EPAD Proof of Concept Trials (with additional consent).
5. Have a study partner or can identify someone willing to be a study partner. The primary role of the study partner will be as informant. They will also receive oral and written information about the EPAD LCS, and will sign an Informed Consent Form (ICF).

Exclusion Criteria:

1. Individuals who fulfill diagnostic criteria for any type of dementia.
2. Clinical Dementia Rating >=1
3. Known carriers of a Presenilin (PSEN) 1, PSEN 2 or Amyloid Precursor Protein (APP) mutation associated with Autosomal Dominant Alzheimer's dementia or any other neurodegenerative disease.
4. Presence of any neurological, psychiatric or medical conditions associated with a long-term risk of significant cognitive impairment or dementia including but not limited to pre- manifest Huntington's disease, multiple sclerosis, Parkinson's disease, Down syndrome, active alcohol/drug abuse; or major psychiatric disorders including current major depressive disorder, schizophrenia, schizoaffective or bipolar disorder.
5. Cancer or history of cancer in the last 5 years (excluding cutaneous basal or squamous cell cancer resolved by excision).
6. Any current medical conditions that are clinically significant and might make participation in an investigational trial unsafe, e.g., uncontrolled or unstable disease of any major organ system; history within the last 6 months of any acute illness of a major organ system requiring emergency care or hospitalization, including revascularization procedures; severe renal or hepatic failure; unstable or poorly controlled DM, hypertension, or heart failure; malignant neoplasms within the last 3 years (expect for basal or squamous cell carcinoma in situ of the skin, or localized prostate cancer in male participants); any clinically relevant abnormalities in blood parameters included in local TDC routine assessments; severe loss of vision, hearing or communicative ability; or any conditions preventing co-operation or completion of the required assessments in the trial, as judged by the investigator.
7. Contraindications for MRI/Positron emission tomography (PET) Scan.
8. Contraindications for Lumbar Puncture.
9. Any evidence of intracranial pathology which, in the opinion of the Investigator, may affect cognition including but not limited to brain tumours (benign or malignant), aneurysm or arteriovenous malformations, territorial stroke (excluding smaller watershed strokes), recent haemorrhage (parenchymal or subdural), or obstructive hydrocephalus. Research participants with a MRI scan demonstrating markers of small vessel disease (e.g. white matter changes or lacunar infarcts) judged to be clinically insignificant, or microbleeds are allowed.
10. Participation in a clinical trial of an Investigational Product (CTIMP) in the last 30 days (continued participation in the parent cohort is expected). Participation in a non-CTIMP is not an exclusion criterion.

Diminished decision-making capacity/ not capable of consenting at Visit 1 or Visit 2. If at a subsequent annual EPAD LCS visit health professionals suspect diminished consent capacity according to local TDC routine procedures, a formal assessment of the research participant's capacity to consent will be conducted. The participant will be offered the opportunity to continue in the EPAD LCS under suitable local regulations regarding capacitous participants who have consented to enter a longitudinal study who subsequently loose capacity. Capacity will be assessed at each study visit using the correct legal framework.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Research participants will mainly be recruited from existing Parent Cohorts (PC) across Europe. PCs considered for EPAD are: active cohorts without dementia aged at least 50 years; the PC PI is willing to provide research participants for EPAD trials; with existing consent for re-contact or possibility to obtain consent to re-contact. Potential research participants will be identified based on data in the PC, using a flexible search algorithm adapted to the types of data available in each PC. Recruitment will be complemented with research participants who are recruited from a clinical setting by their referring clinician. In case an individual or their referring clinician contacts a TDC, the referring clinician will check the flexible algorithm to confirm their suitability.
Sampling Method: Non-Probability Sample
Enrollment: 2095 (Actual)
Dates: Start 2016-05; Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Change in RBANS Composite score over time, units on a scale. | Measured at Baseline, 6 months, year 1, year 2, year 3.
  Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Composite score combining: List Learning & Story Memory; Figure Recall; Figure Copy & Line Orientation; Picture Naming; Semantic Fluency, Digit Span, Coding.

SECONDARY OUTCOMES:
Change in other Secondary Cognitive Tests score: Working Memory, over time, units on a scale. | Measured at Baseline, 6 months, year 1, year 2, year 3
  Dot Counting test
Change in other Secondary Cognitive Tests score: Choice Reaction Time and Set Shifting, over time, units on a scale. | Measured at Baseline, 6 months, year 1, year 2, year 3
  Flanker test
Change in other Secondary Cognitive Tests score: Paired Associate Learning, over time, units on a scale. | Measured at Baseline, 6 months, year 1, year 2, year 3
  Favourites
Change in cerebrospinal fluid (CSF) AD biomarkers over time | Measured at Baseline, year 1, year 2, year 3
  Aβ, t-tau and p-tau levels in pg/ml
Changes in neuro-imaging assessment of hippocampal and whole brain volume, over time | Measured at Baseline, year 1, year 2, year 3
  Hippocampal and whole brain volume, cm3

OTHER OUTCOMES:
Change in exploratory Cognitive Tests score: Allocentric space, over time, units on a scale. | Measured at Baseline, 6 months, year 1, year 2, year 3
  Four Mountains Test
Change in exploratory Cognitive Tests score: Egocentric space, over time, units on a scale. | Measured at Baseline, 6 months, year 1, year 2, year 3
  Supermarket Trolley Virtual Reality Test
Change in other secondary clinical outcome scale: Everyday functioning, total over time, units on a scale | Measured at Baseline, 6 months, year 1, year 2, year 3
  Everyday functioning: Amsterdam Instrumental Activities of Daily Living Questionnaire.
Changes in neuro-imaging assessments over time, Multi-regional Structural and Functional MRI & Functional regional and network measures, units on a scale | Measured at Baseline, year 1, year 2, year 3
  Cortical thickness, deep grey matter (GM) volumes, Fractional anisotropy (FA) of temporal lobe, diffusion kurtosis (multi b-value DTI), network alterations, Global & parietal Cerebral Blood Flow (CBF), Changes within the default-mode network (DMN) & relation with hippocampal activity (rsfMRI), Bolus arrival time (multi-delay ASL), Network analysis (rsfMRI)
Changes in Lifestyle factors over time: Smoking | Measured at Baseline, year 1, year 2, year 3
  Smoking: never/past/current
Changes in Lifestyle factors over time: Alcohol Consumption | Measured at Baseline, year 1, year 2, year 3
  Alcohol: units/week
Changes in Lifestyle factors over time: drug abuse/misuse | Measured at Baseline, year 1, year 2, year 3
  Drug abuse/misuse: never/past/current
Changes in Lifestyle factors over time: diet HATICE (Healthy Aging through Internet Counselling in the Elderly), units on a scale | Measured at Baseline, year 1, year 2, year 3
  Diet questionnaire: HATICE (Healthy Aging through Internet Counselling in the Elderly), physical activity.
Changes in Lifestyle factors over time: physical activity frequency | Measured at Baseline, year 1, year 2, year 3
  Physical activity: daily, 2-3 times/week, 2-3 times/month, a few times a year, not at all
Changes in Lifestyle factors over time: Life events over time | Measured at Baseline, year 1, year 2, year 3
  Life events: SNAC (Swedish National study on Ageing and Care).
Changes in Lifestyle factors over time: Self-rated health and fitness | Measured at Baseline, year 1, year 2, year 3
  Self-rated health and fitness: Very good/good/satisfactory/relatively poor/poor
Change in Mini-Mental Satus Exam (MMSE) over time | Measured at Baseline, year 1, year 2, year 3
  Measure of clinical state
Change in Clinical Dementia Rating Scale (CDR) over time | Measured at Baseline, year 1, year 2, year 3
  Assessment of six domains, (memory, orientation, judgement and problem solving, community affairs, home and hobbies and personal care), from which the global CDR score, CDR sum of notes and a CDR rating for each domain are calculated.
Change in other clinical outcome scale: Depression, total over time, units on a scale | Measured at Baseline, year 1, year 2, year 3
  Depression: Geriatric Depression Scale
Change in other clinical outcome scale: Anxiety, total over time, units on a scale | Measured at Baseline, year 1, year 2, year 3
  Anxiety: State-Trait Anxiety Inventory
Change in other clinical outcome scale: Sleep, total over time, units on a scale | Measured at Baseline, year 1, year 2, year 3
  Sleep: Pittsburgh Sleep Quality Index
Other neuro-imaging measure: Vascular Burden, over time, units on a scale | Measured at Baseline, year 1, year 2, year 3
  Vascular Burden: Counts of White Matter Lesions, infarcts, laciness, micro bleeds and superficial siderosis.
Other clinical outcome: Dementia Diagnosed by a Participant's Physician | Measured at Baseline, year 1, year 2, year 3
  Type of Dementia and Date of Diagnosis
Genetic Assessment of apolipoprotein E (ApoE) genotype | Measured at Baseline
  APOE genotype determined by allele combination of e2, e3 and e4
Sociodemographic Factors (subject to local regulations | Measured at Baseline
  Date of Birth, Age, Ethnicity, Education, Marital Status, Handedness
Other clinical measure: Family History of AD | Measured at Baseline
  Family history of AD in number of family members of first degree with history compatible with AD
Other clinical measure: Medical History | Measured at Baseline, year 1, year 2, year 3
  Medical History: Yes/No for: Stroke, Diabetes (type 1 or 2), Hypertension, Hypercholesterolemia, Myocardial Infarction, Chronic Ischemic Heart Disease, Chronic Obstructive Pulmonary Disease, Asthma, Depression, Rheumatoid Arthritis, Any Cancer, General Anaesthesia after the age of 50 years, Head Injury assessed with the Brain Injury Screening Questionnaire (BISQ), Mild Cognitive Impairment, Other Conditions (Listed as free text)
Other clinical measure: Current Medication | Measured at Baseline, year 1, year 2, year 3
  Drug, treatment duration (<1year / 1-5years / >5years)
Other clinical measure: Body Height | Measured at Baseline
  Body Height: without shoes, measured to the nearest cm
Other clinical measure: Body Weight | Measured at Baseline, year 1, year 2, year 3
  Body Weight: measured to the nearest 0.1kg
Other clinical measure: Hip-waist Circumference | Measured at Baseline, year 1, year 2, year 3
  Hip-waist Circumference: measured to nearest 0.1cm

CONTACTS AND LOCATIONS:
Overall Officials: Craig Ritchie, Principal Investigator — University of Edinburgh
Locations (30):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc ASBL, Neurology Department, Brussels
  - UZ Leuven, Campus Gasthuisberg, Leuven
- France (6):
  - CMRR du CHRU de Lille Hôpital Roger Salengro, Lille
  - CHU Gui de Chauliac Département de Neurologie, Montpellier
  - Groupe Hospitalier Saint Louis - Lariboisière - Fernand Widal, Paris
  - Hôpital Universitaire de la Pitié Salpêtrière, Paris
  - CMRR- Hôpital Laënnec Nord - CIC Neurologie / CHU de Nantes, Saint-Herblain
  - Toulouse University Hospital / Gérontopôle-Research Clinical Center, Toulouse
- National and Kapodistran, University of Athens, 1st Department of Neurology, Aeginition Hospital, Athens, Greece
- Italy (2):
  - Univerita di Perugia, Centro Disturbi della Memoria, Clinica Neurologica, Perugia, Loc. S Andrea Delle Fratte
  - IRCCS San Giovanni di Dio - Fatebenefratelli, Brescia
- VUmc Alzheimer Center and Alzheimer Research Center, Amsterdam, North Holland, Netherlands
- Spain (4):
  - Unidade Deterioro Cognitivo, Servicio de Neurologia, Hospital Universitario, Santander, Cantabria
  - BarcelonaBeta Brain Research Centre, Barcelona
  - Fundacion ACE, Institut Catala de Neurocienies Aplicades, Barcelona
  - Fundacion CITA-alzheimer Fundazioa, Center for Research and Advanced Therapies, San Sebastián
- Sweden (2):
  - Neuropsychiatric Research Unit, Sahlgrenska University Hoospital, Gothenburg, Västra Götaland County
  - Karolinska Institutet, Stockholm
- Switzerland (2):
  - Hôpitaux Universitaires de Genève - HUG, Geneva
  - Centre Leenaards de la memoire- CHUV, Department of Neurosciences cliniques, Lausanne
- United Kingdom (10):
  - Monklands University Hospital, Cumbernauld, Lanarkshire
  - University of Edinburgh, Centre for Dementia Prevention, Edinburgh, Midlothian
  - NHS Grampian, Aberdeen
  - North Bristol NHS Trust, Bristol
  - University of Cambridge; Department of Clinical Neurosciences, Cambridge
  - NHS Tayside, Dundee
  - Glasgow Clinical Research Facility; NHS Greater Glasgow and Clyde, Glasgow
  - West London Mental Health NHS Trust, London
  - Greater Manchester Clinical Research Network, Manchester
  - University of Oxford, Department of Psychiatry, Oxford

IPD SHARING:
Plan to Share IPD: Yes
EPAD is an Innovative Medicines Initiative (IMI) project with open access to data.
Time Frame: Post December 2019
Access Criteria: To be determined by the EPAD Research Access Committee

REFERENCES:
- [Derived] Osset-Malla M, Martinez-Velasco A, Sanchez-Benavides G, Buongiorno M, de la Sierra A, Shekari M, Minguillon C, Kollmorgen G, Quijano-Rubio C, Zetterberg H, Blennow K, Garcia DV, Suarez-Calvet M, Gispert JD, Grau-Rivera O; ALFA Study. Blood pressure and Alzheimer's disease biomarkers in cognitively unimpaired adults: a multicenter study. J Prev Alzheimers Dis. 2025 Dec;12(10):100304. doi: 10.1016/j.tjpad.2025.100304. Epub 2025 Aug 11. PMID 40796457
- [Derived] Vermunt L, Muniz-Terrera G, Ter Meulen L, Veal C, Blennow K, Campbell A, Carrie I, Delrieu J, Fauria K, Huesa Rodriguez G, Ingala S, Jenkins N, Molinuevo JL, Ousset PJ, Porteous D, Prins ND, Solomon A, Tom BD, Zetterberg H, Zwan M, Ritchie CW, Scheltens P, Luscan G, Brookes AJ, Visser PJ; IMI-EPAD collaborators. Prescreening for European Prevention of Alzheimer Dementia (EPAD) trial-ready cohort: impact of AD risk factors and recruitment settings. Alzheimers Res Ther. 2020 Jan 6;12(1):8. doi: 10.1186/s13195-019-0576-y. PMID 31907067
- [Derived] Solomon A, Kivipelto M, Molinuevo JL, Tom B, Ritchie CW; EPAD Consortium. European Prevention of Alzheimer's Dementia Longitudinal Cohort Study (EPAD LCS): study protocol. BMJ Open. 2019 Feb 19;8(12):e021017. doi: 10.1136/bmjopen-2017-021017. PMID 30782589